CLINICAL TRIAL: NCT03307304
Title: Investigations of Juvenile Neuronal Ceroid Lipofuscinosis (CLN3) and CLN3-Related Conditions
Brief Title: Investigations of Juvenile Neuronal Ceroid Lipofuscinosis
Status: Recruiting | Type: Observational
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 180002; 18-CH-0002
Record Dates: First submitted 2017-10-07; First posted 2017-10-11 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01-20

CONDITIONS: Juvenile Neuronal Ceroid Lipofuscinosis (CLN3); Batten Disease
Keywords: Batten Disease; Neurodegenerative; Lysosomal Storage; Biomarkers; Longitudinal Study; Natural History
MeSH Terms: conditions — Neuronal Ceroid-Lipofuscinoses

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Family members: Unaffected family members of individuals diagnosed with CLN3-Batten
- Proband/Affected Individuals: Individuals diagnosed with CLN3-Batten

SUMMARY:
Background:

CLN3, or Batten disease, is a genetic disorder. This deadly disease leads to decline of brain and nervous system functions. Symptoms of CLN3 typically occur between 4 and 7 years of age. They include changes in how a person sees, thinks, and moves. CLN3 can also cause seizures. No effective treatments for the disease are yet known. There is limited testing of potential therapies. Researchers want to study CLN3 more so they can improve future therapies.

Objective:

To identify clinical or biochemical markers that can be used as therapeutic outcome measures for CLN3.

Eligibility:

People with CLN3. It must be based on

Two CLN3 mutations OR

One CLN3 mutation AND findings seen with a powerful microscope

Family members of a person with CLN3.

Design:

Participants will have already been referred to NIH for CLN3 evaluation.

If participants agree to do the study, they will:

1. give spinal fluid, blood, urine, and skin samples. They may provide other samples if they were already collected. These may include cells, surgical specimens, and DNA.
2. will be seen by multiple healthcare specialists.

Participants may provide medical records or photos. Participants will sign a release of medical records form.P

Researchers may send samples or clinical data to other investigators. For research testing, the samples will not include the participant s name. For a test in a clinical lab, researchers will include the participant s name. These results will become part of the clinical record at NIH.

DETAILED DESCRIPTION:
Study Description:

The purpose of this protocol is to obtain both baseline and rate of progression data on clinical and biochemical markers that may later be used as an outcome measure in a clinical trial, and to establish a biorepository of samples from participants with CLN3 or CLN3-

related conditions. For comparisons, focused clinical data and relevant evaluations and biospecimens will also be collected from individuals with Neuronal Ceroids Lipofuscinosis (NCL) of other types and from family members of all affected individuals.

Objectives:

Primary Objective:

1. Identify clinical or biochemical markers that can be used as therapeutic outcome measures for CLN3-related conditions.
2. Evaluate clinical aspects of CLN3-related conditions to provide tools for future therapeutic trials.

Secondary Objectives:

Establish a biorepository of samples from well-characterized individuals with CLN3-related conditions, and family members of individuals with CLN3-related conditions, for future research related to CLN3.

Endpoints:

Primary Endpoint:

1. Blood, urine, or CSF biomarkers.
2. Proportion of participants who achieve a clinically valid and interpretable score on administered measures.
3. Scores obtained for each administered measure.

Secondary Endpoints:

Tolerability and feasibility of each measure of the clinical battery of assessments based on clinician observation.

ELIGIBILITY:
* INCLUSION CRITERIA:

For the Main and Sub-Studies, participants > 1 week of age, of all genders, demographics, geographic locations, and disease severity will be recruited in order to obtain cross-sectional representation of CLN3-related conditions (Main and Sub-Studies) or all NCLs (Sub-Study B). Participants in the Main study will be followed at approximately yearly intervals to obtain longitudinal data. Participants in Sub-Study A may elect to send in medical records and samples only, or to come to the NIH for evaluations as outlined in Section 4. We anticipate that

participants in Sub-Study B will be seen mostly at NCL/CLN3-related family conferences.

Main Study:

Individuals > 1 week of age with a diagnosis of CLN3 or a CLN3-related/other NCL-type condition. Diagnosis determined by one of the following:

1. Two CLN3 or NCL condition-appropriate genetic mutations
2. One CLN3 mutation AND

i) clinical presentation suggestive of CLN3, OR

ii) characteristic electron microscopy (EM) findings (such as curvilinear body, fingerprint profile, granular osmiophilic deposits).

Sub-Study A:

Individuals > 1 week of age with a diagnosis of CLN3 or CLN3-related/other NCL-type condition. Diagnosis determined by one of the following:

1. Two CLN3 or condition-appropriate genetic mutations
2. One CLN3 mutation AND

i) clinical presentation suggestive of CLN3, OR

ii) characteristic electron microscopy (EM) findings (such as curvilinear body, fingerprint profile, granular osmiophilic deposits).

OR

Individuals > 1 month of age who have family member(s) diagnosed with CLN3 or CLN3-related/other NCL-type condition.

Sub-Study B:

Individuals > 1 week of age with a clinical diagnosis of CLN3 or NCL.

OR

Individuals > 1 month of age who have family member(s) diagnosed with CLN3 or NCL.

EXCLUSION CRITERIA:

Main Study:

1. Individuals who cannot travel to the NIH because of their medical condition.
2. Individuals who, in the opinion of the Investigator, are unable to comply with the protocol or have medical conditions that would potentially increase the risk of participation.
3. Females who are pregnant.

Sub-Studies A and B:

1. Unaffected individuals > 18 years of age who have cognitive impairments.
2. Individuals who, in the opinion of the Investigator, are unable to comply with the protocol or have medical conditions that would potentially increase the risk of participation.

Ages: 1 Week to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals with CLN3-Batten and family members who are interested in the study and have consented to enroll.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2017-11-27 (Actual); Primary Completion 2050-12-31 (Estimated); Study Completion 2050-12-31 (Estimated)

PRIMARY OUTCOMES:
Identify clinical or biochemical markers that can be used as a therapeutic outcome measures for CLN3. | ongoing
  Identification of biomarkers
Evaluate clinical aspects of CLN3 to provide tools for future therapeutic trials | ongoing
  Evaluation of clinical signs and symptoms

SECONDARY OUTCOMES:
Establish a biorepository of samples from well-characterized CLN3 patients for future research related to CLN3 | ongoing
  Collection of biospecimens

CONTACTS AND LOCATIONS:
Overall Officials: An N Dang Do, M.D., Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Derived] Luckett A, Yousef M, Tifft C, Jenkins K, Smith A, Munoz A, Quimby R, Porter FD, Dang Do AN. Anesthesia outcomes in lysosomal disorders: CLN3 and GM1 gangliosidosis. Am J Med Genet A. 2023 Mar;191(3):711-717. doi: 10.1002/ajmg.a.63064. Epub 2022 Dec 2. PMID 36461157
- [Derived] Dang Do AN, Thurm AE, Farmer CA, Soldatos AG, Chlebowski CE, O'Reilly JK, Porter FD. Use of the Vineland-3, a measure of adaptive functioning, in CLN3. Am J Med Genet A. 2022 Apr;188(4):1056-1064. doi: 10.1002/ajmg.a.62607. Epub 2021 Dec 16. PMID 34913584
- [Derived] Abdennadher M, Inati S, Soldatos A, Norato G, Baker EH, Thurm A, Bartolini L, Masvekar R, Theodore W, Bielekova B, Porter FD, Dang Do AN. Seizure phenotype in CLN3 disease and its relation to other neurologic outcome measures. J Inherit Metab Dis. 2021 Jul;44(4):1013-1020. doi: 10.1002/jimd.12366. Epub 2021 Feb 15. PMID 33550636
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2018-CH-0002.html